CLINICAL TRIAL: NCT01629316
Title: CID 1007 - Randomized Controlled Trial of an Augmented Test, Treat, Link & Retain Model for NC and TX Prisoners (imPACT Study)
Brief Title: Evaluation of Behavioral Intervention for HIV Positive Prisoners in NC and TX
Acronym: imPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David A Wohl, MD, Clinical Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CID 1007 - UNC IRB 10-1183; R01DA030793-01 (NIH)
Record Dates: First submitted 2012-06-04; First posted 2012-06-27 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: HIV Infection
Keywords: HIV; prisoners; test; treat; link coordination; retain; behavioral; intervention; text reminders; motivational interviewing; medication adherence
MeSH Terms: conditions — HIV Infections; Behavior; Medication Adherence | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Text reminders, counseling, link coordinator (Experimental): Text reminders, counseling, link coordination
  Interventions: Behavioral: Text reminders, counseling, and link coordination
- Standard of care - control arm (Active Comparator)
  Interventions: Behavioral: Standard of care - control arm

INTERVENTIONS:
Behavioral: Text reminders, counseling, and link coordination — This is an intervention with text reminders, counseling that involves motivational interviewing, and link coordination
  Arms: Text reminders, counseling, link coordinator
Behavioral: Standard of care - control arm — The control arm is standard of care for each subject.
  Arms: Standard of care - control arm

SUMMARY:
Purpose: The purpose of this study is to determine if a comprehensive intervention supporting seek-test-and-treat results in a significant reduction in the potential for HIV-infected prisoners to transmit their virus after release from prison.

Aim 2: Compare the effect of standard prison test-and-treat (sTNT) with the TNT-imPACT (imPACT) intervention on viral load 24 weeks following prison release.

Aim 3: Describe and model secondary outcomes, comparing them between sTNT and TNT-imPACT study arms. These outcomes include post-release HIV transmission risk behaviors, incident STIs, adherence to ART, medical care appointments, emergence of ART resistance mutations, and predicted HIV transmission events.

DETAILED DESCRIPTION:
For Aims 2 and 3:

Participants:

We will enroll 400 HIV-infected men and women, age 18 years and older who are incarcerated in the NC Department of Correction (NCDOC) or the Texas Department of Criminal Justice (TDCJ) and scheduled for prison release in approximately 12 weeks, who are receiving ART and have an HIV RNA level that is below 400 copies/mL.

Procedures (methods): Participants will be consented, enrolled, and then randomized 1:1 to one of two conditions:

1. standard test-and-treat (sTNT), which is the current standard of care, wherein following HIV testing, the DOC provides to HIV-infected inmates ART during incarceration and referral to community-based care and services by prison staff as well as a supply of antiretroviral medication (30 days in NC, 10 in TX) upon release, or
2. TNT-imPACT (imPACT),which includes the sTNT plus our integrated, multi-component intervention targeting multiple levels to enhance adherence to HIV therapy and linkage to and engagement in clinical care, to maintain viral suppression after release.

All participants will be followed for up to 24 weeks post-release.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Incarcerated in the NCDOC at a facility within a 3 hour drive from Chapel Hill OR incarcerated in the TDCJ at a facility within a 3 hour drive from Ft. Worth
* Age 18 years or older
* Receiving ART for at least 30 days
* Last recorded viral load (must be within 90 days of entry) <400 copies/mL
* English speaking
* Able and willing to provide informed consent
* Willing to participate in post-release study activities
* For NC - planning to remain in state after release and returning to a community within a 3 hour drive of Chapel Hill
* For TX - returning to one of the following areas: Houston, Dallas, and Ft. Worth (including their suburbs)
* Scheduled for release from prison

Exclusion Criteria:

* Conviction for offenses that includes sexual assault or death or serious injury to a victim or is otherwise found, in the opinion of the investigators, to be at high risk for injury to staff (this criterion is designed to minimize risk to study personnel who will conduct study-related visits with participants in the communities to which they return and may be informed by input from correctional staff)
* Pending charges that would likely lead to transfer of custody or other condition which would otherwise prevent or significantly delay release from custody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2012-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
HIV RNA level (Viral Load) | Week 24 post-release from prison

CONTACTS AND LOCATIONS:
Overall Officials: David A Wohl, MD, Principal Investigator — University of North Carolina, Chapel Hill; Carol Golin, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Texas Christian University, Fort Worth, Texas

REFERENCES:
- [Background] Granich RM, Gilks CF, Dye C, De Cock KM, Williams BG. Universal voluntary HIV testing with immediate antiretroviral therapy as a strategy for elimination of HIV transmission: a mathematical model. Lancet. 2009 Jan 3;373(9657):48-57. doi: 10.1016/S0140-6736(08)61697-9. Epub 2008 Nov 27. PMID 19038438
- [Background] Lima VD, Johnston K, Hogg RS, Levy AR, Harrigan PR, Anema A, Montaner JS. Expanded access to highly active antiretroviral therapy: a potentially powerful strategy to curb the growth of the HIV epidemic. J Infect Dis. 2008 Jul 1;198(1):59-67. doi: 10.1086/588673. PMID 18498241
- [Background] Dieffenbach CW, Fauci AS. Universal voluntary testing and treatment for prevention of HIV transmission. JAMA. 2009 Jun 10;301(22):2380-2. doi: 10.1001/jama.2009.828. No abstract available. PMID 19509386
- [Background] Spaulding AC, Seals RM, Page MJ, Brzozowski AK, Rhodes W, Hammett TM. HIV/AIDS among inmates of and releasees from US correctional facilities, 2006: declining share of epidemic but persistent public health opportunity. PLoS One. 2009 Nov 11;4(11):e7558. doi: 10.1371/journal.pone.0007558. PMID 19907649
- [Background] Leukefeld CG, Staton M, Hiller ML, Logan TK, Warner B, Shaw K, Purvis RT. A descriptive profile of health problems, health services utilization, and HIV serostatus among incarcerated male drug abusers. J Behav Health Serv Res. 2002 May;29(2):167-75. doi: 10.1007/BF02287703. PMID 12032974
- [Background] Springer SA, Pesanti E, Hodges J, Macura T, Doros G, Altice FL. Effectiveness of antiretroviral therapy among HIV-infected prisoners: reincarceration and the lack of sustained benefit after release to the community. Clin Infect Dis. 2004 Jun 15;38(12):1754-60. doi: 10.1086/421392. Epub 2004 May 26. PMID 15227623
- [Background] Baillargeon J, Giordano TP, Rich JD, Wu ZH, Wells K, Pollock BH, Paar DP. Accessing antiretroviral therapy following release from prison. JAMA. 2009 Feb 25;301(8):848-57. doi: 10.1001/jama.2009.202. PMID 19244192
- [Background] Stephenson BL, Wohl DA, Golin CE, Tien HC, Stewart P, Kaplan AH. Effect of release from prison and re-incarceration on the viral loads of HIV-infected individuals. Public Health Rep. 2005 Jan-Feb;120(1):84-8. doi: 10.1177/003335490512000114. PMID 15736336
- [Background] Haley D, Scheyett A, Golin C, et al. Perceptions of Release among Incarcerated HIV-Infected Persons and Implications for Practice: The UNC Bridges to Good Health and Treatment (BRIGHT) Project Qualitative Substudy. Abstract THPE0717. International AIDS Conference, 2006
- [Background] Stephenson BL, Wohl DA, McKaig R, Golin CE, Shain L, Adamian M, Emrick C, Strauss RP, Fogel C, Kaplan AH. Sexual behaviours of HIV-seropositive men and women following release from prison. Int J STD AIDS. 2006 Feb;17(2):103-8. doi: 10.1258/095646206775455775. PMID 16464271
- [Background] Grinstead O, Zack B, Faigeles B. Reducing postrelease risk behavior among HIV seropositive prison inmates: the health promotion program. AIDS Educ Prev. 2001 Apr;13(2):109-19. doi: 10.1521/aeap.13.2.109.19737. PMID 11398956
- [Background] Best A, Stokols D, Green LW, Leischow S, Holmes B, Buchholz K. An integrative framework for community partnering to translate theory into effective health promotion strategy. Am J Health Promot. 2003 Nov-Dec;18(2):168-76. doi: 10.4278/0890-1171-18.2.168. PMID 14621414
- [Background] Stokols D. Translating social ecological theory into guidelines for community health promotion. Am J Health Promot. 1996 Mar-Apr;10(4):282-98. doi: 10.4278/0890-1171-10.4.282. PMID 10159709
- [Derived] Golin CE, Knight K, Carda-Auten J, Gould M, Groves J, L White B, Bradley-Bull S, Amola K, Fray N, Rosen DL, Mugavaro MJ, Pence BW, Flynn PM, Wohl D. Individuals motivated to participate in adherence, care and treatment (imPACT): development of a multi-component intervention to help HIV-infected recently incarcerated individuals link and adhere to HIV care. BMC Public Health. 2016 Sep 6;16(1):935. doi: 10.1186/s12889-016-3511-1. PMID 27596559
- See also: Maruschak LM, Beavers R. Bureau of justice statistics: HIV in prisons, 2007-08. U.S. Department of Justice: Bureau of Justice Statistics; 2009 12/09. Report No.: NCJ 228307. http://bjs.ojp.usdoj.gov/content/pub/pdf/hivp08.pdf — http://bjs.ojp.usdoj.gov/content/pub/pdf/hivp08.pdf
- See also: 15. Sabol WJ, West H and Cooper M. Bureau of justice statistics: Prisoners in 2008. U.S. Department of Justice: Bureau of Justice Statistics; 2009 12/09. Report No.: NCJ 228417. http://bjs.ojp.usdoj.gov/index.cfm?ty=pbdetail&iid=1763 — http://bjs.ojp.usdoj.gov/index.cfm?ty=pbdetail&iid=1763